CLINICAL TRIAL: NCT01505387
Title: Double-blind, Randomized, Placebo-controlled Clinical Investigation to Evaluate the Safety and Efficacy of Litramine in Maintaining Body Weight Loss in Overweight and Obese Subjects
Brief Title: Litramine in Weight Maintenance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ/024511
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Weight Maintenance; Overweight; Obese
Keywords: Weight maintenance; Overweight; Obese; Weight management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Identical to Litramine 2 tablets 3 times daily (oral consumption, after meal)
  Interventions: Dietary Supplement: Placebo
- Litramine (Experimental): Fibre complex of plant origin n tablet form 2 tablets 3 times daily (oral consumption, after meal)
  Interventions: Dietary Supplement: Litramine

INTERVENTIONS:
Dietary Supplement: Litramine — Fibre complex of plant origin in tablet form 2 tablets 3 times daily (oral consumption, after meal)
  Arms: Litramine
Dietary Supplement: Placebo — Identical to Litramine tablets 2 tablets 3 times daily (oral consumption, after meal)
  Arms: Placebo

SUMMARY:
The effect of Litramine on weight loss has previously been studied during a 12-week intervention period with promising results. The present study looks into the effect of weight maintenance using Litramine following initial weight loss, for a longer period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented weight loss, achieved over the last 3 to 6 months either from participation in weight loss clinical trials or weight loss regimens, of at least 3% at the point of screening
* BMI 25-35 before initial weight loss
* Documented compliance (according to the investigator's judgement) to previous weight loss clinical trials/ regimens

Exclusion Criteria:

* Known sensitivity to the ingredients of the device (citric acid, acacia or Fabaceae family)
* BMI < 18.5
* Presence of other factor(s) that, in the investigator's judgement, should preclude subject participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Grube, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Grube B, Chong PW, Alt F, Uebelhack R. Weight Maintenance with Litramine (IQP-G-002AS): A 24-Week Double-Blind, Randomized, Placebo-Controlled Study. J Obes. 2015;2015:953138. doi: 10.1155/2015/953138. Epub 2015 Sep 7. PMID 26435849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial conducted from January 2012 to September 2012 in two study sites in Germany
Period: Overall Study
Arm/Group | Placebo | Litramine
Started | 25 | 25
Treated | 24 | 24
Completed | 23 (1 subject not included in intention to treat population as violated inclusion criteria) | 24
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Litramine | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.2) | 44.7 (11.4) | 44.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 6 | 6 | 12
Body weight (kg) [Mean (Standard Deviation); unit: kg] | 79.3 (9.0) | 78.2 (11.4) | 78.7 (10.2)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (2.4) | 27.3 (2.1) | 27.5 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Body Weight From Baseline to End of 24 Weeks
Description: Change in body weight at the end of 24 weeks measured in kg using a calibrated scale. (positive values signify weight gain, while negative values signify weight reduction
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Litramine
Number analyzed (Participants) | 24 | 25
kg | 1.62 (1.48) | -0.62 (1.55)

2. Secondary Outcome: Waist and Hip Circumference (cm)
Description: Changes from baseline to end of study
Time Frame: 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Body Mass Index (kg/m^2)
Description: Changes from baseline to end of study
Time Frame: 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Full Blood Count
Description: Erythrocytes, leukocytes, thrombocytes, haematocrit, haemoglobin, Mean corpuscular volume (MCV), Mean corpuscular haemaglobin (MCH)
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Blood Pressure
Description: Measured in mm Hg
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Litramine
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other